CLINICAL TRIAL: NCT04056130
Title: A Phase I Randomized Double-blind Placebo-controlled Study of Single and Multiple Ascending Doses of KBL697 in Healthy Subjects
Brief Title: A Study of Single and Multiple Ascending Doses of KBL697 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KoBioLabs (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KBL-CURE-2019-01
Record Dates: First submitted 2019-07-24; First posted 2019-08-14 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort SAD1 (Experimental): 9 Subjects for SAD 1 Cohort. 6 subjects on KBL697, 3 subjects on Placebo.
  Interventions: Drug: KBL697
- Cohort SAD2 (Experimental): 9 Subjects for SAD 2 Cohort. 6 subjects on KBL697, 3 subjects on Placebo.
  Interventions: Drug: KBL697
- Cohort MAD1 (Experimental): 9 Subjects for MAD 1 Cohort. 6 subjects on KBL697, 3 subjects on Placebo
  Interventions: Drug: KBL697
- Cohort MAD2 (Experimental): 9 Subjects for MAD 2 Cohort. 6 subjects on KBL697, 3 subjects on Placebo
  Interventions: Drug: KBL697

INTERVENTIONS:
Drug: KBL697 — Part A: 1 day 460mg/day of KBL697 or placebo
  Route of Administration: Oral
  Other Names: Placebo
  Arms: Cohort SAD1
Drug: KBL697 — Part A: 1 day 4,600mg/day of KBL697
  Route of Administration: Oral
  Other Names: Placebo
  Arms: Cohort SAD2
Drug: KBL697 — Part B: 14 days
  Cohort MAD1:
  460mg/day of KBL697
  Route of Administration: Oral
  Other Names: Placebo
  Arms: Cohort MAD1
Drug: KBL697 — Part B: 14 days
  Cohort MAD2:
  4,600mg/day of KBL697
  Route of Administration: Oral
  Other Names: Placebo
  Arms: Cohort MAD2

SUMMARY:
The study is designed to investigate the safety and tolerability of KBL697 in healthy volunteers. KBL697 has been developed as a potential new treatment for atopic dermatitis (AD).

DETAILED DESCRIPTION:
This is a randomized double-blind, placebo-controlled, single centre Phase I study.

Thirty-six (36) subjects are planned to be randomised at

1 site across the 2 parts of the study as follows:

* Part A (Single Ascending Dose (SAD) in healthy subjects)
* Part B (Multiple Ascending Doses (MAD) in healthy subjects)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able to read and understand, and willing to sign the informed consent form (ICF)
2. Male or female, aged 18 to 60 years (inclusive) at the time of Screening
3. Body mass index (BMI) of 18 kg/m2 to ≤ 30 kg/m2 (both inclusive)
4. Willing and able to comply with clinic visits (including confinement to clinical trial unit) and study-related procedures
5. No history of allergic asthma
6. Baseline laboratory test values within reference ranges based on the blood and urine samples taken at screening and on Day -1. Out of normal ranges values may be accepted by the Investigator, if not clinically significant.
7. Male subjects must abstain from heterosexual activities or agree to use a condom from screening through 90 days after the final dose of study drug. Women of child-bearing potential (WOCBP) must also abstain from heterosexual activities or agree to use effective contraception from screening through 90 days after the final dose of study drug.
8. Ability to remain in the study centre for up to a 3-day period for Part A of the study and up to a 15-day period for Part B of the study.
9. The subject is, in the opinion of the Investigator, generally healthy based on assessment of medical history, physical examination, vital signs, electrocardiogram (ECG), and the results of the haematology, clinical chemistry, urinalysis, serology, and other relevant laboratory tests.
10. Subject willing to allow storage of samples for genetic make-up in future studies.

Exclusion Criteria:

1. Female participants who are pregnant or lactating
2. The participant's corrected QT interval (QTcF) (Fridericia's correction) is >450 msec (males), and >470 msec (females) at Screening or on Day -1. An out-of-range or abnormal ECG will be repeated at PI's discretion. In total, 3 ECGs should be recorded consecutively at Screening and on Day -1, and the PI (or delegate) must evaluate the triplicate ECG. If the participant's QTcF is >450 msec (males) or >470 msec (females) on at least 2 ECGs or have structural cardiac abnormalities, the participant must be excluded
3. The participant has taken prescription (including antibiotics) or non-prescription medication, herbal remedies, vitamins or minerals, any probiotic drinks and yeast supplements (e.g. Mutaflor®, Bioflor®) within 14 days prior to the first dose of study product unless in the opinion of the PI the medication will not compromise participant safety or interfere with study procedures or data validity. Participant may be rescreened after a washout period of 14 days. Please note use of oral contraceptives and paracetamol up to 2 g/day and/or nonsteroidal anti-inflammatory drugs for symptomatic relief of minor symptoms are allowed
4. Participant has functional GI disorders
5. Participant is a current smoker or has used nicotine containing products within 6 months prior to Screening visit
6. The participant has a substance abuse-related disorder or has a history of drug, alcohol and/or substance abuse deemed significant by the PI
7. The participant has taken any IP within 30 days prior to the first dose of study product or 5 half-lives, whichever is longer
8. The participant has a history of significant hypersensitivity or anaphylaxis involving any drug (including ampicillin, clindamycin or imipenem), any constituent of the IP, food or other precipitating agent (e.g. bee sting). Please note participants with clinically stable mild allergic conditions such as hay fever and mild eczema may be enrolled at the discretion of the PI
9. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus antibody (anti-HCV)at Screening visit.
10. Positive screen for drugs of abuse and cotinine at Screening or on Day -1. Positive screen for alcohol on Day -1.
11. The participant is, in the opinion of the PI, unlikely to comply with the clinical study protocol or is unsuitable for any other reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability measure through Adverse Events/Serious Adverse Events | Measurements at Baseline till 28 days
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Safety and tolerability measure through Vital Sign | Measurement at Baseline till 28 days
  Measured by result of the Vital Sign(blood pressure, heart rate, axillary body temperature, respiratory rate)
Safety and tolerability measure through 12-lead ECG | Measurement at Baseline till 28 days
  Measured by result of the ECG measurements and findings
Safety and tolerability measure through Physical exam | Measurement at Baseline till 28 days
  Measured by result of the physical exam which includes general appearance, skin, eyes/ears/nose/throat, head and neck, cardiovascular, respiratory, abdomen, extremities, lymph nodes, musculoskeletal and neurologic
Safety and tolerability measure through Routine Stool Examination | Measurement at Baseline till 28 days
  Measured by result of the Bristol Stool Examination, Occult blood, Parasites
Safety and tolerability measure through Clinical laboratory results | Measurement at Baseline till 28 days
  Measured by clinically significant change from baseline clinical laboratory results

OTHER OUTCOMES:
Difference in the change from baseline in profile of faecal KBL697 between treatment arms | Measurements at Baseline till 28 days
  Measured by quantitative analysis method for understanding distribution and excretion of KBL697

CONTACTS AND LOCATIONS:
Overall Officials: Ben Snyder, Dr, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No